CLINICAL TRIAL: NCT05354583
Title: Comparison Study of Unfavorable Treatment Outcome Between Mycobacterium Abscessus Infection in Patients With Chronic Lung Disease and Acquired Interferon-gamma Autoantibody Syndrome Within 1 Year of Appropriate Treatment
Brief Title: Treatment Outcome Between Mycobacterium Abscessus Infection in Chronic Lung Disease and Acquired Interferon-gamma Autoantibody Syndrome
Status: Completed | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Warat Usawakidwiree, Internal medicine resident, King Chulalongkorn Memorial Hospital
Other Study IDs: 46/2565
Record Dates: First submitted 2022-04-06; First posted 2022-04-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Mycobacterium Abscessus Infection; Adult-Onset Immunodeficiency With Acquired Anti-Interferon-Gamma Autoantibodies; Nontuberculous Mycobacterial Pulmonary Infection
Keywords: Mycobacterium Abscessus Infection; Adult-Onset Immunodeficiency with Acquired Anti-Interferon-Gamma Autoantibodies; Nontuberculous Mycobacterial Pulmonary Infection
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acquired Interferon-gamma Autoantibody Syndrome: Patients infected with M. abscessus at any site, who have acquired interferon-gamma autoantibody syndrome defined as one of the following features:
  1. The M. abscessus infection site is lymph node.
  2. The M. abscessus infection is disseminated (more than 1 organ of infection or blood culture positive for M. abscessus).
  3. The M. abscessus infection is accompanied by one of reactive skin diseases which are Sweet's syndrome, pustular psoriasis, erythema nodosum.
  4. History of opportunistic infection such as salmonellosis, penicillosis, histoplasmosis, cryptococcosis, melioidosis
  The patients must not be infected with HIV, in-hospital M. abscessus infection, diagnosed with cancer, or receiving immunosuppressants.
  Interventions: Drug: Appropriate treatment
- Chronic Lung Disease: Patients with one of chronic lung diseases which are COPD, chronic bronchiectasis, history of pulmonary tuberculosis and diagnosed with Pulmonary M. abscessus infection.
  Pulmonary M. abscessus infection diagnosis must be met all of the following criteria:
  1. Symptoms and signs are correlated with the pulmonary M. abscessus infection.
  2. One of the radiological evidences:
     2.1) nodular infiltration or cavitary lesion on plain chest radiography
     2.2) bronchiectasis and multiple small nodules on chest computerized tomography
  3. Mycobacterial culture from respiratory tract specimen is positive for M. abscessus
  Interventions: Drug: Appropriate treatment

INTERVENTIONS:
Drug: Appropriate treatment — Treatment with at least 3 antibiotics, which the pathogen is susceptible to based on in vitro drug susceptibility test, in the initial phase of the treatment

SUMMARY:
The treatment outcome of Mycobacterium abscessus infection in acquired interferon-gamma autoantibody syndrome has not been well studied. Investigators will perform a retrospective and prospective cohort study to determine the treatment outcome of Mycobacterium abscessus infection in patients with acquired interferon-gamma autoantibody syndrome compared with the infection in patients with chronic lung disease which is known to be the most common group of infection and have high rates of treatment failure. Investigators hypothesized that Mycobacterium abscessus infection in acquired interferon-gamma autoantibody syndrome has better outcome than infection in chronic lung disease.

DETAILED DESCRIPTION:
The single center, retrospective and prospective cohort study including the patients, aged 18 years and over, with acquired interferon-gamma autoantibody syndrome or chronic lung disease diagnosed with M. abscessus infection in the tertiary hospital of Thailand from January 2014 to June 2023 will be perform. The enrolled M. abscessus infected patients will be divided into two groups which are acquired interferon-gamma autoantibody syndrome group and chronic lung disease group. The subjects' medical record will be reviewed for demographic data, underlying diseases, clinical signs and symptoms, laboratory and radiological investigation results, diagnosis, treatment that the patients received, clinical events during the treatment. The treatment outcome will be determined as unfavorable or favorable by present or absent of unfavorable events, settled by the investigators, within 1 years after the treatment. The treatment outcome and other secondary outcomes between the two groups will then be compared and analysed with chi-squared test for categorical variables and two-sample t-test for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Diagnosed with Mycobacterium abscessus pulmonary disease in chronic lung disease or Mycobacterium abscessus infection in acquired interferon-gamma autoantibody syndrome
* Receive appropriate treatment

Exclusion Criteria:

* Follow up time less than one year after the start of appropriate treatment
* Very incomplete medical record that the subject's history cannot be reviewed
* Appropriate treatment duration less than one year at the study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit King Chulalongkorn Memorial Hospital (a tertiary care hospital in Thailand) during the study period
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Unfavorable Treatment Outcome | The start of appropriate treatment to one year after that
  The occurring of any unfavorable events including
  1. Clinical unfavorable events which are 1.1) death relating to M. abscessus infection 1.2) ongoing or worsening of symptoms or signs of infection after 6 weeks of treatment 1.3) addition new class or changing class of antibiotics during treatment (not included changing antibiotics according to in vitro susceptibility test)
  2. Radiological unfavorable event which is stable or worsen radiological features related to M. abscessus infection after 6 weeks of treatment
  3. Microbiological unfavorable events which are 3.1) Acid fast bacilli positive from clinical specimen after 6 weeks of treatment 3.2) Mycobacterial culture positive for M. abscessus after 6 weeks of treatment

SECONDARY OUTCOMES:
Demographic data | At the time that M. abscessus infection is diagnosed through study completion, about one year
  Age, sex, nationality, religion, occupation, birth place, current residence
Proportion of Subspecies of Mycobacterium abscessus | At the time that M. abscessus infection is diagnosed through study completion, about one year
  Subspecies from the first mycobacterial culture result including subsp. abscessus, massiliense, and boletii
Drug resistance rate of Mycobacterium abscessus | At the time that M. abscessus infection is diagnosed through study completion, about one year
  Rate of resistance to each class of antibiotics acquired from the first in vitro susceptibility test that is done as resisted, susceptible, or intermediate

CONTACTS AND LOCATIONS:
Overall Officials: Warat Usawakidwiree, M.D., Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand; Chusana Suankratay, M.D., Ph.D., Study Director — Division of Infectious Diseases, Department of Internal Medicine, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand